CLINICAL TRIAL: NCT01186666
Title: BIOmarkers of CORonary Events-2 : Imaging and Biomarkers of Atherosclerosis in Patients With Stable or Unstable Coronary Artery Disease
Brief Title: Imaging and Biomarkers of Atherosclerosis in Patients With Stable or Unstable Coronary Artery Disease
Acronym: BIOCORE-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P080703
Record Dates: First submitted 2010-07-12; First posted 2010-08-23 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Atherosclerosis; Coronary Artery Disease; Acute Coronary Syndrome
Keywords: Atherosclerosis; Vulnerable plaque; Intravascular ultrasound; Virtual histology; Fluorodeoxyglucose; Positron emission tomography; Multidetector computed tomography
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non ST-elevation acute coronary syndrome (Experimental): Coronary intervention using IVUS-VH & FDG PET-MDCT:
  All the patients will undergo percutaneous coronary intervention of culprit vessels after imaging of the entire coronary tree (culprit and non-culprit lesions) using intravascular ultrasound with radiofrequency data analysis (IVUS-VH). Before discharge, fluorodeoxyglucose positron emission tomography combined with multidetector computed tomography (FDG PET-MDCT) of the carotid arteries and the thoracic aorta, along with MDCT coronary angiography, will be performed and a blood sample will be obtained for subsequent measurements of emerging or new biomarkers.
  Interventions: Device: Coronary intervention using IVUS-VH & FDG PET-MDCT
- Stable coronary artery disease (Experimental): Coronary intervention using IVUS-VH & FDG PET-MDCT:
  All the patients will undergo percutaneous coronary intervention of culprit vessels after imaging of the entire coronary tree (culprit and non-culprit lesions) using intravascular ultrasound with radiofrequency data analysis (IVUS-VH). Before discharge, fluorodeoxyglucose positron emission tomography combined with multidetector computed tomography (FDG PET-MDCT) of the carotid arteries and the thoracic aorta, along with MDCT coronary angiography, will be performed and a blood sample will be obtained for subsequent measurements of emerging or new biomarkers.
  Interventions: Device: Coronary intervention using IVUS-VH & FDG PET-MDCT

INTERVENTIONS:
Device: Coronary intervention using IVUS-VH & FDG PET-MDCT — All the patients will undergo percutaneous coronary intervention of culprit vessels after imaging of the entire coronary tree (culprit and non-culprit lesions) using intravascular ultrasound with radiofrequency data analysis (IVUS-VH). Before discharge, fluorodeoxyglucose positron emission tomography combined with multidetector computed tomography (FDG PET-MDCT) of the carotid arteries and the thoracic aorta, along with MDCT coronary angiography, will be performed and a blood sample will be obtained for subsequent measurements of emerging or new biomarkers.
  Arms: Non ST-elevation acute coronary syndrome
Device: Coronary intervention using IVUS-VH & FDG PET-MDCT — All the patients will undergo percutaneous coronary intervention of culprit vessels after imaging of the entire coronary tree (culprit and non-culprit lesions) using intravascular ultrasound with radiofrequency data analysis (IVUS-VH). Before discharge, fluorodeoxyglucose positron emission tomography combined with multidetector computed tomography (FDG PET-MDCT) of the carotid arteries and the thoracic aorta, along with MDCT coronary angiography, will be performed and a blood sample will be obtained for subsequent measurements of emerging or new biomarkers.
  Arms: Stable coronary artery disease

SUMMARY:
In this study, multimodal imaging of atherosclerosis and dosage of new circulating biomarkers will be used to compare patients with stable or unstable coronary artery disease

DETAILED DESCRIPTION:
Acute complications of coronary and cerebrovascular atherosclerosis -i.e., acute coronary syndromes (ACS) and strokes - remain the principal cause of death worldwide. Identification of patients at high risk of developing such complications is therefore of utmost importance. Post-MORTEM studies suggest that vulnerable coronary atherosclerotic plaques are characterized by a large, metabolically active, necrotic core, covered by a thin fibrous cap, which may rupture, leading to acute thrombosis, myocardial infarction and, potentially, sudden death. These anatomic features of plaque vulnerability are not visible on standard coronary imaging, such as coronary angiography, but might be recognized using more recent imaging modalities. In addition, new circulating biomarkers of atherosclerosis, particularly biomarkers involved in plaque destabilization, can be measured in peripheral blood and may be used to appreciate overall patient vulnerability.

Design and Methods- In the present study, 2 groups of 44 patients with moderate-to-high risk non-ST elevation ACS or stable coronary artery disease (CAD) will be compared. All the patients will undergo percutaneous coronary intervention of culprit vessels after imaging of the entire coronary tree (culprit and non-culprit lesions) using intravascular ultrasound with radiofrequency data analysis (IVUS-VH). Before discharge, fluorodeoxyglucose positron emission tomography combined with multidetector computed tomography (FDG PET-MDCT) of the carotid arteries and the thoracic aorta, along with MDCT coronary angiography, will be performed and a blood sample will be obtained for subsequent measurements of emerging or new biomarkers.

Objectives -

1. The primary objective is to compare plaque phenotypes between patients with ACS vs stable CAD. For each imaging modality (coronary IVUS-VH, MDCT coronary angiography, AORTO-carotid FDG PET-CT) comparisons will be performed on a per-lesion and per-patient basis.
2. Secondary objectives include: i) An evaluation of the accuracy of each plaque imaging modality and biomarkers for diagnosis of unstable CAD; ii) A comparison of the diagnostic performance of each plaque imaging modality and biomarkers for diagnosis of unstable CAD; iii) A comparison of coronary plaque phenotype between culprit and non-culprit lesions (using IVUS-VH and MDCT coronary angiography); and iv) An exploratory feasibility study of PET-CT imaging of coronary artery atherosclerotic plaques.

It's important to underline that this study must be considered as an interventional study. Indeed, in this study patients have many imaging modality : coronary IVUS-VH, MDCT coronary angiography and AORTO-carotid FDG PET-CT while in common practice patients have only FDG PET-CT which is the routinely technique used.

ELIGIBILITY:
Inclusion Criteria:

First group: Non ST-elevation acute coronary syndrome

* Symptoms compatible with acute myocardial ischaemia
* Presence of either significant ST-T changes without persistent ST elevation or positive troponin I
* And successful stenting of culprit, de novo coronary stenosis located on native coronary arteries

Second group: Stable coronary artery disease

* Stable angina or silent myocardial ischaemia (documented by a positive stress test)
* And successful stenting of culprit, de novo coronary stenosis located on native coronary arteries

Exclusion Criteria:

In both groups

* Absence of percutaneous coronary angioplasty
* IVUS imaging not feasible
* Heart failure (≥NYHA class 2)
* Severe, persistent arrhythmia
* Renal failure (GFR < 60 ml/min using MDRD formula)
* History of autoimmune or inflammatory disease, recent sepsis (< 1 month), neoplasm
* Females without contraception (if at childbearing age)
* Pregnant of child feeding females
* Homeless
* Patients with no health coverage
* Refusal to sing informed consent
* Allergy to FDG or iodinated contrast media

In stable group:

* History of acute coronary syndrome
* History of stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-02; Primary Completion 2012-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Three imaging modalities are used to compare plaque phenotypes between patients with ACS vs stable CAD. (coronary IVUS-VH, MDCT coronary angiography, AORTO-carotid FDG PET-CT) | Performed within 7 days of inclusion
  Each imaging modality provides a set of quantitative or semi-quantitative measures of plaque vulnerability (eg, necrotic core volume and presence of thin-cap fibroatheroma on IVUS-VH; presence of calcium and positive remodeling on MDCT coronary angiography; and FDG uptake measured by target-to-background on aorto-carotid FDG PET-CT)

SECONDARY OUTCOMES:
New circulating biomarkers | Measured on a blood sample performed within 7 days of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Feldman, MD, PhD, Study Director — Assistance Publique Hopitaux de Paris
Locations (1):
- Département de Cardiologie, Hôpital Bichat, Assistance Publique - Hôpitaux de Paris, Paris, France

REFERENCES:
- [Derived] Loyau S, Dumont B, Ollivier V, Boulaftali Y, Feldman L, Ajzenberg N, Jandrot-Perrus M. Platelet glycoprotein VI dimerization, an active process inducing receptor competence, is an indicator of platelet reactivity. Arterioscler Thromb Vasc Biol. 2012 Mar;32(3):778-85. doi: 10.1161/ATVBAHA.111.241067. Epub 2011 Dec 8. PMID 22155453